CLINICAL TRIAL: NCT01625104
Title: Randomized Trial of Aggressive Process of Care Quality Improvement Intervention to Decrease Door to Balloon Time in Primary PCI for Acute Myocardial Infarction
Brief Title: Randomized Trial of a Quality Improvement Intervention to Decrease D2B Time in Primary PCI for AMI
Acronym: RAPID-PCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Blue Cross Blue Shield of Michigan Foundation (Other)
Responsible Party: Principal Investigator, Eva Kline-Rogers, Study Coordinator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1998-0080
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Results first posted 2017-12-15 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-05

CONDITIONS: STEMI
Keywords: Myocardial Infarction; Time to Treatment; Door to Balloon Time
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: Aggressive Intervention Strategy (Experimental): Hospitals were randomized to an aggressive intervention strategy or to "business as usual". The hospitals randomized to the aggressive intervention strategy underwent the following:
  1. Grand Rounds conducted by physician and nurse from the Coordinating Center. This included a formal presentation on the evidence supporting rapid time to treatment in STEMI patients and evidence based strategies for reducing treatment delays.
  2. Discussion with staff regarding perceived barriers to treatment and suggestions/ideas for strategies to overcome these barriers
  3. Follow-up monthly phone conferences to continue to discuss strategies and ideas sharing
  4. Written plan from sites detailing plans to change processes of care.
  Interventions: Other: Agressive Intervention Process Improvement Strategies
- Group 2: Control Strategy (Placebo Comparator): Hospitals randomized to the control group were instructed to conduct "business as usual".
  Interventions: Other: Non Intervention

INTERVENTIONS:
Other: Non Intervention — Business as usual
  Arms: Group 2: Control Strategy
Other: Agressive Intervention Process Improvement Strategies
  Arms: Group 1: Aggressive Intervention Strategy

SUMMARY:
The primary objective of this study is to assess whether an aggressive quality improvement intervention strategy will decrease time from hospital presentation to first balloon inflation in non-transfer patients with acute ST segment elevation MI (STEMI) treated with primary percutaneous coronary intervention (PCI). Twelve hospitals in Michigan were randomized to either aggressive intervention or control. The intervention consisted of Grand Rounds at each hospital, sharing of best practices, and coordinating center staff working closely with staff at each intervention hospital to discuss solutions to barriers to rapid treatment for STEMI patients.

DETAILED DESCRIPTION:
The participating hospitals randomized to the aggressive intervention strategy actively worked to create teams to analyze processes of care for STEMI patients, identify areas needing improvement, and implemented strategies to streamline treatment.

Hospitals randomized to control were instructed to conduct "business as usual".

ELIGIBILITY:
Inclusion Criteria:

* Acute ST segment myocardial infarction, non transfer patients, with symptom onset to balloon time less than or equal to 24 hours.

Exclusion Criteria:

* Patients transferred from one facility to another,
* non ST segment myocardial infarction patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 882 (Actual)
Dates: Start 2003-09; Primary Completion 2006-02 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Moscucci, M.D., Principal Investigator — University of Michigan; Eva M Kline-Rogers, MS, RN, Study Director — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 6 sites were randomized to the aggressive strategy and 6 sites were randomized to control.
Pre-assignment Details: Site were randomized according to baseline Door to Balloon times.
Groups:
- Group 1: Agressive Strategy: Hospitals were randomized to an aggressive intervention strategy or to "business as usual". The hospitals randomized to the aggressive intervention strategy underwent the following:
  1. Grand Rounds conducted by physician and nurse from the Coordinating Center. This included a formal presentation on the evidence supporting rapid time to treatment in STEMI patients and evidence based strategies for reducing treatment delays.
  2. Discussion with staff regarding perceived barriers to treatment and suggestions/ideas for strategies to overcome these barriers
  3. Follow-up monthly phone conferences to continue to discuss strategies and ideas sharing
  4. Written plan from sites detailing plans to change processes of care.
- Group 2: Control: Hospitals randomized to the control group were instructed to conduct "business as usual".
Period: Overall Study
Arm/Group | Group 1: Agressive Strategy | Group 2: Control
Started | 448 | 434
Completed | 448 | 434
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Agressive Intervention: Hospitals were randomized to an aggressive intervention strategy or to "business as usual". The hospitals randomized to the aggressive intervention strategy underwent the following:
  1. Grand Rounds conducted by physician and nurse from the Coordinating Center. This included a formal presentation on the evidence supporting rapid time to treatment in STEMI patients and evidence based strategies for reducing treatment delays.
  2. Discussion with staff regarding perceived barriers to treatment and suggestions/ideas for strategies to overcome these barriers
  3. Follow-up monthly phone conferences to continue to discuss strategies and ideas sharing
  4. Written plan from sites detailing plans to change processes of care.
- Group 2: Control Strategy: Hospitals randomized to the control group were instructed to conduct "business as usual".
  Business as usual was described as site specific protocol for treatment of STEMI patient +/- any ongoing quality improvement efforts. No specific recommendations were given to sites from the coordinating center.
- Total: Total of all reporting groups
Arm/Group | Group 1: Agressive Intervention | Group 2: Control Strategy | Total
Number analyzed (Participants) | 448 | 434 | 882
Age, Continuous [Median (Standard Deviation); unit: years] | 61.2 (13.2) | 60.2 (12.4) | 60.7 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 134 | 270
  Male | 312 | 300 | 612

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Sites With Reduction in Door to Balloon Time
Description: Arrival time in Emergency Department to first balloon inflation in the coronary artery.
  Any reduction in median Door to Balloon Time from baseline to follow-up was counted as reduction in time
Time Frame: Arrival to balloon inflation, measured in minutes (generally less than 120 mins)
Measure: Number; unit: percentage of sites with improved D2B
Arm/Group | Group 1: Aggressive Stategy | Group 2: Control Strategy
Number analyzed (Participants) | 448 | 434
percentage of sites with improved D2B | 83 | 50

ADVERSE EVENTS:
Groups:
- Group 2: Control Strategy: Hospitals randomized to the control group were instructed to conduct "business as usual".
  Business as usual was defined as normal protocol for treatment of STEMI patients at each individual site +/- quality improvement efforts. No contact or advice was given to the sites from the coordinating center.
Arm/Group | Group 1: Agressive Intervention | Group 2: Control Strategy
Serious Adverse Events (participants affected / at risk) | 0/448 | 0/434
Other Adverse Events (participants affected / at risk) | 0/448 | 0/434

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No